CLINICAL TRIAL: NCT00788346
Title: Reducing Unnecessary Use of Heavily Marketed Medicines: A Randomized Controlled Trial of Computerized Prescribing Alerts and Clinician Education
Brief Title: Reducing the Unnecessary Use of Heavily Marketed Medications: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Oregon (Other)
Responsible Party: Steven R. Simon, MD (Principal Investigator), Harvard Medical School and Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5.12.05
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2008-11

CONDITIONS: Use of Sleep Medications
Keywords: Heavily marketed medications; Prescribing; Health information technology; Education
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Computerized Alerts (Experimental): Computerized Clinical Decision Support to clinician at the time of prescribing
  Interventions: Behavioral: Computerized alerts
- Alerts PLUS Detailing (Experimental): Computerized Clinical Decision Support to clinician at the time of prescribing PLUS one group academic detailing session
  Interventions: Behavioral: Alerts Plus Detailing
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Computerized alerts — Computerized Clinical Decision Support to clinician at the time of prescribing
  Arms: Computerized Alerts
Behavioral: Alerts Plus Detailing — Computerized Clinical Decision Support to clinician at the time of prescribing PLUS one group academic detailing session
  Arms: Alerts PLUS Detailing

SUMMARY:
Prescribing decisions by clinicians are often thought to be simple: a patient's clinical problem leads a prescriber to choose the optimal treatment. However, many factors other than the patient's condition affect prescribing decisions, including the marketing of pharmaceuticals. Clinicians are subjected to direct "detailing" by representatives of the pharmaceutical industry, advertisements in medical journals and requests for specific treatments from patients, who are increasingly exposed to direct-to-consumer (DTC) advertising. These influences, often based on biased or inaccurate information, contribute to a variety of problems in prescribing, including the unnecessary use of expensive, heavily marketed medications.

Overcoming these influences requires innovative approaches. The movement toward widespread adoption of electronic health records (EHRs) and electronic prescribing presents new opportunities to educate both clinicians and patients at the time of medication prescribing. This project, endorsed by the AHRQ-supported Centers for Education and Research on Therapeutics (CERTs; www.certs.hhs.gov) and the U.S. Food and Drug Administration (FDA), aims to test the effectiveness of computerized prescribing alerts and state-of-the-art educational outreach to reduce the unnecessary use of heavily marketed medications. A second goal is to improve clinicians' knowledge of industry marketing practices, so that they can more effectively assess information provided by drug companies. Thus, the study has two specific aims:

Specific Aim 1: To assess whether computerized prescribing alerts linked electronically to patient educational material can reduce prescribing of heavily marketed medications.

Specific Aim 2: To assess whether group academic detailing increases clinicians' knowledge about industry marketing practices and increases the effect of prescribing alerts.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine clinicians

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
proportion of prescriptions for hypnotic medications that were heavily marketed medications (study medications). Hypnotic medications were defined as the study medications intervention plus zolpidem and trazodone. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Simon, MD, Principal Investigator — Harvard Medical School and Harvard Pilgrim Health Care
Locations (1):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fortuna RJ, Zhang F, Ross-Degnan D, Campion FX, Finkelstein JA, Kotch JB, Feldstein AC, Smith DH, Simon SR. Reducing the prescribing of heavily marketed medications: a randomized controlled trial. J Gen Intern Med. 2009 Aug;24(8):897-903. doi: 10.1007/s11606-009-1013-x. Epub 2009 May 28. PMID 19475459